CLINICAL TRIAL: NCT03781115
Title: Proposal To Develop A Rapid And Cost-Effective Diagnostic Test For Schizophrenia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Sidney R. Baer, Jr. Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1612051594
Record Dates: First submitted 2017-10-13; First posted 2018-12-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: schizophrenia, psychosis, ziprasidone, olanzapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — ziprasidone; Olanzapine

STUDY DESIGN:
Intervention Model Description: The investigators will first conduct a dose-response evaluation of the anti-psychotic drug ziprasidone (Geodon) (20, 40, or 60 mg tablet) or olanzapine (Zyprexa®) (2.5, 5, 7.5, or 10 mg tablet) in non-psychiatric ill control individuals to determine the dosage that promotes sedation in individuals versus a placebo. The evaluation will comprise a physical examination, drug/pregnancy screenings and sleepiness questionnaires. Once the dosage of the anti-psychotic medication is determined new healthy subjects will be recruited to ingest the medication and have an electroencephalogram (EEG) recording taken. If the dosage of medication does not show an effect on the EEG the investigators will ask the individual to come back on a different day so the next higher dose of medication can be given. Once a the healthy subject's EEG shows an effect new control subjects and individuals with a diagnosis of schizophrenia will be recruited.
Who Masked: Participant, Investigator
Masking Description: Double Blind Masking: The participant and the investigator are both blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ziprasidone (Experimental): The investigators will conduct a pilot dose-response evaluation of a single dose of the anti-psychotic drug ziprasidone (Geodon). The investigators will start with a single 20mg pill given to (3) subjects and will increase the dosage in sequential subjects until the desired sedation effect is achieved (i.e. 40 and 60mg tablets). If Ziprasidone causes the desired sedation effect additional healthy subjects will be recruited to take the medication and have an electroencephalogram (EEG) taken.
  Interventions: Drug: Ziprasidone; Drug: Olanzapine; Drug: Placebo Comparator
- Olanzapine (Experimental): The investigators will conduct a pilot dose-response evaluation of a single dose of the anti-psychotic drug olanzapine (Zyprexa). The investigators will start with a single 2.5 mg pill given to (3) subjects and will increase the dosage in sequential subjects until the desired sedation effect is achieved (i.e. 5, 7.5, and 10 mg tablets).If olanzapine causes the desired sedation effect additional healthy subjects will be recruited to take the medication and have an electroencephalogram (EEG).
  Interventions: Drug: Olanzapine; Drug: Placebo Comparator
- Placebo Comparator (Placebo Comparator): The investigators have prepared a placebo which duplicates the exact color and size of the study drug capsule to use as a non-drug control.
  Interventions: Drug: Ziprasidone; Drug: Placebo Comparator

INTERVENTIONS:
Drug: Ziprasidone — anti-psychotic drug proposed for use as rapid diagnostic tool
  Other Names: Geodon
  Arms: Placebo Comparator; Ziprasidone
Drug: Olanzapine — anti-psychotic drug proposed for use as rapid diagnostic tool
  Other Names: Zyprexa
  Arms: Olanzapine; Ziprasidone
Drug: Placebo Comparator — A non drug oral placebo capsule will be given as a control
  Other Names: Placebo Oral Capsule

SUMMARY:
Schizophrenia is a severe psychotic illness of unknown cause that affects 1% of the population worldwide. Currently, there is no diagnostic test for schizophrenia. Instead, the diagnosis is typically established through a psychiatric interview of the patient, who is evaluated against a set of established criteria of signs and symptoms. It can take many months to years to establish a diagnosis of schizophrenia and achieve an appropriate treatment regimen to attain resolution of the patient's symptoms. This process is particularly challenging in areas of limited access to specialists a problem not only in third world countries and rural regions, but throughout the United States where there can be long waits to obtain an appointment with a psychiatrist. The present research experiment investigates a potential novel method for diagnosing schizophrenia.

The overall objective of the study is to test the hypothesis that patients with schizophrenia will have a heightened tolerance to the sedating effects of anti-psychotic medications, which will be reflected in differences in their electroencephalogram (EEG) when compared to healthy normal controls. The investigators expect that the schizophrenia patients will score on the "more alert" and "less sleepy" ends of these scales, and that the normal control subjects will show the opposite response. A patient that fails to become sedated or experience the sleepiness side effects, typically caused by the anti-psychotic medication, may support the existing diagnosis of schizophrenia. Measures of the subjects' level of sedation that are found to correlate significantly with EEG response and diagnosis will be used to create a diagnostic test. This simple and inexpensive test will consist of a single dosage of anti-psychotic medication, and a rapid assessment tool with scores that have a high degree of predictive validity for the diagnosis of schizophrenia.

DETAILED DESCRIPTION:
The overall objective of the study is to test the hypothesis that patients with schizophrenia will have a heightened tolerance to the sedating effects of antipsychotic medications, which will be reflected in differences in the participants' electroencephalogram response (EEG), when compared to healthy control participants.The following Specific Aims are designed to test this hypothesis and create the diagnostic tool.

Specific Aim 1: The investigators will first conduct a pilot dose-response evaluation of the anti-psychotic drugs ziprasidone (Geodon) (20, 40, or 60 mg tablet) and olanzapine (Zyprexa®) (2.5, 5, 7.5, or 10 mg tablet) in non-psychiatric ill control participants to determine the optimal dosage that promotes sedation in healthy participants versus a placebo. The evaluation will comprise a physical examination and questionnaires. The investigators will start with the lowest dose of each drug and if the dosage fails to induce sedation in healthy participants, the investigators will repeat the pilot dose-response evaluation with the next higher dose until the maximum dose is reached for both drugs. Specific Aim 2. To determine whether the pattern of EEG activity in response to a single dose of the anti-psychotic medication determined from the dose-response study from Aim 1 distinguishes schizophrenia participants from normal controls. The investigators will start with 2-4 healthy control participants to determine that the results show a discernible effect on the EEG using the dosage from Aim 1. If the dose of anti-psychotic medication fails to show an effect on the EEG the investigators will increase the dosage until the maximum dosage of the chosen medication is used. Once the dosage is identified the investigators will move onto getting IRB approval to evaluate participants diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria Healthy Control

1. Be between 18 and 40 years of age
2. Be able to understand English
3. Have no history of psychosis
4. Have no history of sleep apnea, heart condition or seizure
5. Have no known drug allergies
6. The ability to swallow a pill

Exclusion Criteria Healthy control

1. Refuse to sign the consent form
2. Drink caffeine or alcohol within 24 hours of the study
3. Have the EKG readout report borderline or abnormal ECG
4. Have the 12 panel urine drug screen show a positive result
5. Be pregnant

Inclusion Criteria Schizophrenic subject

1. Be between 18 and 40 years of age
2. Be able to understand English
3. Have been diagnosed with a Schizophrenia Spectrum or other psychotic disorder
4. Belong to one of three groups:

   1. Never medicated patients with a first episode of psychosis
   2. Have not received long acting injectable (depot) antipsychotic in previous 6 months
   3. Have not received oral antipsychotic (or antidepressant that has serotonergic action) in previous 2 weeks
5. Have no history of sleep apnea, heart condition or seizure
6. Have no known drug allergies
7. Be able to swallow a pill
8. Healthy as determined by the enrolling physician(s)

Exclusion Criteria Schizophrenic subject

1. Refuse to sign the consent form
2. Drink caffeine or alcohol within 24 hours of the study
3. Have the EKG readout report borderline or abnormal ECG
4. Have the 12 panel urine drug screen show a positive result
5. Be pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Heart Rate | up to 2 years
  Evaluating the heart rate of the subject every hour during all the test procedures
Pulse Rate | up to 2 years
  Evaluating the pulse rate of the subject every hour during all the test procedures
Stanford Sleepiness Scale | up to 2 years
  The subject will rate how sleepy they are feeling at baseline and every hour during the test using an (8) point scale (i.e. 1= feeling active, vital alert, or wide awake; 2= functioning at high levels, but not fully alert; 3= awake, but relaxed, responsive but not fully alert; 4= somewhat foggy, let down; 5= foggy, losing interest in remaining awake, slowed down; 6= sleepy, woozy, fighting sleep, prefer to lay down; 7= no longer fighting sleep, sleep onset soon, having dream-like thoughts; 8= asleep
Epworth Sleepiness Scale | up to 2 years
  The subject will rate their pre-test sleepiness only once during the test using a (4) point scale (0= no chance of dosing, 1= slight chance of dosing, 2= moderate chance of dozing and 3= high chance of dozing
Fatigue Severity Scale | up to 2 years
  The subject will rate their pre-test fatigue only once during the test by rating 10 questions using a slide scale between 1 and 7. A rating of 1 means the subject strongly disagrees with the statement. A rating of 7 means the subject strongly agrees with the statement.
Chalder Fatigue Scale | up to 2 years
  Subjects will rate their fatigue every hour and at baseline by answering 11 questions and rating their fatigue using a 4 point scale (i.e. less than usual, no more than usual, more than usual and much more than usual)
Psychomotor physical computerized test | up to 2 years
  The participants uses a computerized test to test their reflexes every hour and at baseline during the trial period. Every time a red dot appears in the middle of the screen the participant must touch the computer screen as fast as they can. This test was measured in how fast they responded (ms) and by how many attempts to touch the screen were recorded in 2 minutes
Hand Fatigue Scale | up to 2 years
  A hand grip measuring device will be used to test for fatigue. A small hand held device will measure the participants hand grip strength every hour during the test and at baseline.
Electroencephalogram | up to 2 years
  Electroencephalogram will be taken at baseline and after subjects have taken the anti-psychotic medication. There will be no placebo taken for this test.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Gallitano, MD,PhD, Principal Investigator — University of Arizona College of Medicine
Locations (1):
- Banner University Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cutler NR. Pharmacokinetic studies of antipsychotics in healthy volunteers versus patients. J Clin Psychiatry. 2001;62 Suppl 5:10-3; discussion 23-4. PMID 11305842
- [Background] Gallitano-Mendel A, Izumi Y, Tokuda K, Zorumski CF, Howell MP, Muglia LJ, Wozniak DF, Milbrandt J. The immediate early gene early growth response gene 3 mediates adaptation to stress and novelty. Neuroscience. 2007 Sep 7;148(3):633-43. doi: 10.1016/j.neuroscience.2007.05.050. Epub 2007 Aug 9. PMID 17692471
- [Background] Gallitano-Mendel A, Wozniak DF, Pehek EA, Milbrandt J. Mice lacking the immediate early gene Egr3 respond to the anti-aggressive effects of clozapine yet are relatively resistant to its sedating effects. Neuropsychopharmacology. 2008 May;33(6):1266-75. doi: 10.1038/sj.npp.1301505. Epub 2007 Jul 18. PMID 17637609
- [Background] Williams AA, Ingram WM, Levine S, Resnik J, Kamel CM, Lish JR, Elizalde DI, Janowski SA, Shoker J, Kozlenkov A, Gonzalez-Maeso J, Gallitano AL. Reduced levels of serotonin 2A receptors underlie resistance of Egr3-deficient mice to locomotor suppression by clozapine. Neuropsychopharmacology. 2012 Sep;37(10):2285-98. doi: 10.1038/npp.2012.81. Epub 2012 Jun 13. PMID 22692564
- [Background] Selvaraj S, Arnone D, Cappai A, Howes O. Alterations in the serotonin system in schizophrenia: a systematic review and meta-analysis of postmortem and molecular imaging studies. Neurosci Biobehav Rev. 2014 Sep;45:233-45. doi: 10.1016/j.neubiorev.2014.06.005. Epub 2014 Jun 24. PMID 24971825
- [Background] Everson G, Lasseter KC, Anderson KE, Bauer LA, Carithens RL Jr, Wilner KD, Johnson A, Anziano RJ, Smolarek TA, Turncliff RZ. The pharmacokinetics of ziprasidone in subjects with normal and impaired hepatic function. Br J Clin Pharmacol. 2000;49 Suppl 1(Suppl 1):21S-26S. doi: 10.1046/j.1365-2125.2000.00149.x. PMID 10771450
- [Background] Albaugh VL, Singareddy R, Mauger D, Lynch CJ. A double blind, placebo-controlled, randomized crossover study of the acute metabolic effects of olanzapine in healthy volunteers. PLoS One. 2011;6(8):e22662. doi: 10.1371/journal.pone.0022662. Epub 2011 Aug 9. PMID 21857944